CLINICAL TRIAL: NCT00926952
Title: Safety and Efficacy of Photodynamic Therapy With Short Incubation Methylaminolevulinate Without Occlusion in the Treatment of Actinic Keratoses.
Brief Title: Short Incubation Methylaminolevulinate Photodynamic Therapy Without Occlusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Galderma Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inno-6010
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Results first posted 2011-02-17 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratoses; actinic keratosis; methylamonolevulinate; photodynamic therapy; without occlusion; short incubation
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MAL-PDT 90 min incubation, no occlusion (Experimental): Patients had 2-4 g of Methylaminolevulinate (MAL) spread on the entire face without occlusion and waited 90 minutes prior to photodynamic therapy (PDT) using red light.
  Interventions: Drug: Methylaminolevulinate (Metvix, Metvixia); Device: Photodynamic Therapy (Aktilite)

INTERVENTIONS:
Drug: Methylaminolevulinate (Metvix, Metvixia) — 2-4 g of cream applied to entire face at Day 0 for 90 minutes without occlusion prior to light treatment. If any actinic keratoses remained after 4 weeks the treatment was repeated at Week 4.
  Other Names: Metvix, Metvixia
Device: Photodynamic Therapy (Aktilite) — Device set to 37 J/cm². Red light wavelength is approximately 630 nm.
  Other Names: Aktilite

SUMMARY:
Actinic keratoses on the face are often numerous and widespread. The application of Methylaminolevulinate (MAL) on individual lesions followed by the application of a plastic film on each lesion is difficult and takes time for subjects with many actinic keratoses. The waiting period of 3 hours between MAL cream application and red light exposure is also long for patients. The goal of this study is to evaluate the safety and efficacy of photodynamic therapy (PDT) with MAL with a shorter cream application time (90 minutes) and when MAL is applied on the entire face without the plastic film.

DETAILED DESCRIPTION:
A total of 20 patients with at least 5 non-hypertrophic actinic keratoses (AK) of the face were included in this open-label study. All AKs were mapped on a transparent template before the first PDT treatment. At Day 0, all patients received methylaminolevulinate (MAL) applied on the entire face (except the nose and peri-ocular area of 1-2 cm) without any skin preparation. One to two 2 g MAL tubes was used for the entire face. MAL was applied without occlusion. After a total of 90 +/- 5 minutes the skin was rinsed and exposed to 37 J/cm² of red light from an Aktilite™ device. Patients were seen at Week 4; if all facial AKs did not show a complete response to treatment, the MAL-PDT procedure was repeated at Week 4. Patients were seen again at Week 12 and 24.

The primary endpoint was at Week 12. Patients came back at Week 24 for a final safety evaluation and to verify the recurrence of AK.

Efficacy is evaluated by assessing the mean number of facial AK at Week 12 as compared to Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Patient with at least 5 actinic keratoses of the face at Day 0.
* Patient was willing to use an adequate contraceptive method or was surgically sterile, post menopausal, abstinent or with a same sex partner. Adequate means of contraception included oral contraceptives, IUD in use for 30 days before Day 0, barrier methods and spermicide in use at least 14 days before Day 0.
* Patient capable of giving informed consent.

Exclusion Criteria:

* Patient with allergy to methylaminolevulinate or any component of the vehicle which includes peanut and almond oil.
* Patient with clinically significant sensitivity to visible light, porphyria or porphyrin sensitivity.
* Patient used any topical treatment for actinic keratoses (including imiquimod and 5-fluouracil), on the face within 4 weeks preceding Day 0.
* Patient had cryotherapy or surgery on the face within 4 weeks preceding Day 0.
* Patient with any malignant skin lesion (such as basal cell carcinoma, invasive squamous cell carcinoma or Bowen's disease) on the face at Day 0.
* Patient used photodynamic therapy, with any topical or systemic photosensitizer within 8 weeks preceding Day 0.
* Patient was exposed to excessive ultraviolet radiation (UVB phototherapy, sun tanning salons) within the 4 weeks preceding Day 0.
* Patient used any investigational drug within 4 weeks preceding Day 0.
* Patient with problems of alcoholism or drug abuse in the past year.
* Patient with any unstable or serious uncontrolled medical condition.
* Current pregnancy or lactation.
* Patient with any serious dermatological disorder, including malignancies that would either put the patient at risk or interfere with efficacy or safety evaluations.
* Patient with Fitzpatrick phototype IV, V or VI (inadequate penetration of red light in dark skinned subjects.
* Patients with extensive facial hair (e.g., beard) that would either impair red light exposure or interfere with lesion evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research
Locations (1):
- Innovaderm Research Inc, Montreal, Quebec, Canada

REFERENCES:
- [Background] Griffiths CE, Wang TS, Hamilton TA, Voorhees JJ, Ellis CN. A photonumeric scale for the assessment of cutaneous photodamage. Arch Dermatol. 1992 Mar;128(3):347-51. PMID 1550366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period lasted from July 30, 2009 to July 14, 2010. Type of location was a medical research clinic.
Groups:
- MAL-PDT 90 Min Incubation, no Occlusion: Patients have 2-4 g of Methylaminolevulinate (MAL) spread on the entire face without occlusion and wait 90 minutes prior to photodynamic therapy (PDT) using red light.
Period: Overall Study
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 65.25 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  Canada | 20
Mean Number of Actinic Keratosis lesions on face [Mean (Standard Deviation); unit: Lesions] | 9.85 (7.88)
Mean Griffiths Photonumeric Scale for Photodamage Score [Mean (Standard Deviation); unit: Units on a scale.] — Griffiths photonumeric scale was evaluated by the dermatologist. Patients were placed under natural daylight or fluorescent lighting for grading. A direct comparison was then made between the subjects and photographic standards (provided in reference 1). If an exact match could not be made to a grade then an inter-grade number was used used, for example 1, 3, 5, or 7. Zero (0) is the least amount of photodamage, 8 is the most amount of photodamage.
  Units on a scale. | 5.40 (1.60)
Descriptive Scale -Mean Fine Wrinkling [Mean (Standard Deviation); unit: Units on a scale] — This factor represents a visual assessment of the number and depth of superficial wrinkles (i.e. shallow indentations or lines). Fine wrinkles typically appear in periorbital and perioral regions and are usually found further from the eyes and mouth than are coarse wrinkles.
  * Rating Category
  * 0 None
  * 1-3 Mild
  * 4-6 Moderate
  * 7-9 Severe
  Units on a scale | 5.40 (1.76)
Descriptive Scale - Mean Coarse Wrinkling [Mean (Standard Deviation); unit: Units on a scale] — This factor represents a visual assessment of the number and depth of coarse wrinkles (i.e. deep lines, furrows, or creases). Coarse wrinkles appear on the forehead, glabella, chin, and nasolabial and periorbital areas, and they tend to be located closer to the eyes and mouth than fine wrinkles.
  * Rating Category
  * 0 None
  * 1-3 Mild
  * 4-6 Moderate
  * 7-9 Severe
  Units on a scale | 5.00 (2.20)
Descriptive Scale - Mean Sallowness [Mean (Standard Deviation); unit: Units on a scale] — This factor represents a visual assessment of color tone from very pink or rosy (0) to very sallow or pale (9).
  * Rating Category
  * 0 None
  * 1-3 Mild
  * 4-6 Moderate
  * 7-9 Severe
  Units on a scale | 3.60 (2.37)
Descriptive Scale - Mean Mottled Hyperpigmentation [Mean (Standard Deviation); unit: Units on a scale] — This factor represents a visual assessment of light, patchy, mottled hyperpigmentation and solar freckling (including melasma) based on quantitative criteria such as the area/density of pigment, color intensity (dark vs. light), and uniformity of distribution (i.e. the more uneven or blotchy, the greater the score), Lentigines, nevi, and other pigmented lesions are not to be included in this assessment.
  * Rating Category
  * 0 None
  * 1-3 Mild
  * 4-6 Moderate
  * 7-9 Severe
  Units on a scale | 4.45 (2.14)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Facial Actinic Keratoses at Week 12
Time Frame: 12 weeks
Population: The analysis was per protocol (PP). Imputation techniques were not required since all patients completed the study and no visits were missed.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Lesions | 2.70 (2.32)

2. Secondary Outcome: Number of Patients With Complete Clinical Response of All Actinic Keratoses at Week 12
Description: The proportion of patients with a complete clinical response is calculated by dividing the number of patients with a complete response at week 12 by the number of participants at baseline.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Participants | 3

3. Secondary Outcome: Number of Actinic Keratosis Lesions With Complete Clinical Response at Day 0 and Week 12
Time Frame: 0, 12 weeks
Measure: Number; unit: Lesions
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Lesions
  Day 0 - Total lesions at baseline | 197
  Week 12 - Lesions with complete clinical response | 143

4. Secondary Outcome: Mean Griffiths Photonumeric Scale for Photodamage Score at Week 12
Description: Griffiths photonumeric scale was evaluated by the dermatologist. Patients were placed under natural daylight or fluorescent lighting for grading. A direct comparison was then made between the subjects and photographic standards (provided in reference 1). If an exact match could not be made to a grade then an inter-grade number was used used, for example 1, 3, 5, or 7. Zero (0) is the least amount of photodamage, 8 is the most amount of photodamage.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Units on a scale | 4.85 (1.66)

5. Secondary Outcome: Mean Fine Wrinkling Score at Week 12
Description: This factor represents a visual assessment of the number and depth of superficial wrinkles (i.e. shallow indentations or lines). Fine wrinkles typically appear in periorbital and perioral regions and are usually found further from the eyes and mouth than are coarse wrinkles.
  Rating Category 0 None 1-3 Mild 4-6 Moderate 7-9 Severe
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Units on a scale | 4.30 (1.42)

6. Secondary Outcome: Mean Coarse Wrinkling Score at Week 12
Description: This factor represents a visual assessment of the number and depth of coarse wrinkles (i.e. deep lines, furrows, or creases). Coarse wrinkles appear on the forehead, glabella, chin, and nasolabial and periorbital areas, and they tend to be located closer to the eyes and mouth than fine wrinkles.
  Rating Category 0 None 1-3 Mild 4-6 Moderate 7-9 Severe
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Units on a scale | 4.55 (2.42)

7. Secondary Outcome: Mean Sallowness Score at Week 12
Description: This factor represents a visual assessment of color tone from very pink or rosy (0) to very sallow or pale (9).
  Rating Category 0 None 1-3 Mild 4-6 Moderate 7-9 Severe
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Units on a scale | 3.10 (2.34)

8. Secondary Outcome: Mean Mottled Hyperpigmentation at Week 12
Description: This factor represents a visual assessment of light, patchy, mottled hyperpigmentation and solar freckling (including melasma) based on quantitative criteria such as the area/density of pigment, color intensity (dark vs. light), and uniformity of distribution (i.e. the more uneven or blotchy, the greater the score), Lentigines, nevi, and other pigmented lesions are not to be included in this assessment.
  Rating Category 0 None 1-3 Mild 4-6 Moderate 7-9 Severe
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Units on a scale | 4.40 (1.64)

9. Secondary Outcome: Number of Adverse Events
Description: To study the safety of MAL-PDT performed without occlusion when red light exposure takes place 90 minutes after the application of MAL by tracking adverse events until week 12 and adverse events until week 24
Time Frame: 12, 24 weeks
Population: as for outcome 1
Measure: Number; unit: Adverse events
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Number analyzed (Participants) | 20
Adverse events
  Week 12 | 11
  Week 24 | 0

ADVERSE EVENTS:
Arm/Group | MAL-PDT 90 Min Incubation, no Occlusion
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAL-PDT 90 Min Incubation, no Occlusion (N=20)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAL-PDT 90 Min Incubation, no Occlusion (N=20)
Burning sensation on forehead (Skin and subcutaneous tissue disorders) | 1 (1)
Vitreous detachment left eye (Eye disorders) | 1 (1)
Common Cold (Infections and infestations) | 3 (3)
Erythema application site (General disorders) | 19 (19)
Crusting application site (General disorders) | 1 (1)
Squamous cell carcinoma face (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes